CLINICAL TRIAL: NCT01761617
Title: Yoga Dosing Study for Chronic Low Back Pain in a Predominantly Low-Income Minority Population
Brief Title: Yoga Dosing Study for Chronic Low Back Pain
Acronym: YLBP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AT005956-01A1 (NIH)
Record Dates: First submitted 2012-12-04; First posted 2013-01-07 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2013-01

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Yoga; Chronic Low Back Pain; CAM; Complementary and Alternative Medicine; Minorities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga Class Twice Per Week (Active Comparator): Participants attend two hatha yoga classes each week for 12 weeks.
  Interventions: Behavioral: Yoga class twice per week
- Yoga Class Once per Week (Active Comparator): Participants attend one hatha yoga class each week for 12 weeks.
  Interventions: Behavioral: Yoga class once per week

INTERVENTIONS:
Behavioral: Yoga class once per week — The protocol consists of one 75-minute yoga class per week for 12 weeks. The 12 weeks are divided into four 3-week segments, each with a theme (e.g., "Listening to the Wisdom of the Body," "Engaging your Power"). The number of postures learned and degree of difficulty increases with each segment. The protocol provides variations and uses various aids (e.g., chair, yoga strap, yoga block) to accommodate a range of physical abilities. Classes are taught by a team of yoga instructors to ensure a low participant-to-teacher ratio.
  Arms: Yoga Class Once per Week
Behavioral: Yoga class twice per week — The protocol consists of two 75-minute yoga classes per week for 12 weeks. The 12 weeks are divided into four 3-week segments, each with a theme (e.g., "Listening to the Wisdom of the Body," "Engaging your Power"). The number of postures learned and degree of difficulty increases with each segment. The protocol provides variations and uses various aids (e.g., chair, yoga strap, yoga block) to accommodate a range of physical abilities. Classes will have eight participants at a time and are taught by a team of two yoga instructors to ensure a low yoga participant-to-teacher ratio.
  Arms: Yoga Class Twice Per Week

SUMMARY:
A 12-week randomized controlled trial (RCT) for chronic low back pain in predominantly minority populations comparing yoga classes once/week vs. twice/week. Primary outcomes are pain intensity and measure of disability; secondary outcomes are pain medication use, treatment adherence, and health-related quality of life.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) affects 5-10% of U.S. adults annually and costs over $50 billion per year in direct health care expenditures. Individuals from low-income minority backgrounds are disproportionately impacted by CLBP due to disparities in access and treatment. Several recent studies suggest yoga is effective for CLBP. Yoga may also have other relevant benefits for CLBP patients, such as improved mood, stress reduction, and lower cost. However, there are no studies which directly compare different doses of yoga for CLBP. It is unknown if there is a meaningful dose- response effect of yoga for CLBP. If there is a dose/response effect, the magnitude of the effect is unknown. The total dose of a yoga intervention depends upon the duration of total intervention, frequency of yoga classes, duration of each yoga class, and home practice (amount, duration and frequency).

To assess the impact of yoga dose, we propose conducting a Pilot Yoga Dosing Study for 96 adults from Boston Medical Center. The Dosing Study will be a 12-week randomized controlled trial where participants are assigned to either once per week 75-minute yoga classes or twice per week 75 minute yoga classes.

During this 12-week study, there will be three points of data collection (baseline, 6 weeks, 12 weeks). In addition, little is known about the reliability of different forms of survey administration in low back pain trials. For example, it is unknown if telephone administered questionnaires or web-based data collection are reliable compared to the traditional paper- administered questionnaire.Therefore we will compare different methods of survey administration at each time point. The results of this Pilot will inform the design of a larger future comparative effectiveness RCT of yoga, physical therapy, and education for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Current non-specific low back pain persisting >12 weeks. Mean low back pain intensity for the previous week 4 or greater on a 0 to 10 numerical rating scale (0=no pain to 10=worst possible pain).
* English fluency sufficient to follow treatment instructions and answer survey questions
* Willingness to list comprehensive contact information for at least one (preferably two) friend, family member, or work colleague who will always know how to contact the participant.

Exclusion Criteria:

* Use of yoga in the previous 6 months
* New CLBP treatments started within the previous month or anticipated to begin in the next 12 months
* Pregnancy
* Back surgery in the previous three years
* Specific CLBP pathologies
* Severe or progressive neurological deficits
* Sciatica pain equal to or greater than back pain
* Active substance or alcohol abuse
* Active or planned worker's compensation, disability, or personal injury claims

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Average pain intensity | up to 12 weeks
  Measured on 0-10 scale; asked at baseline, 6 weeks and 12 weeks
Modified Roland Morris Disability Questionnaire for back pain-specific disability | up to 12 weeks
  Roland Morris Disability Questionnaire is a widely used health status measure for low back pain; asked at baseline, 6 weeks and 12 weeks

SECONDARY OUTCOMES:
Pain medication use | up to 12 weeks
  Asked at baseline, 6 weeks and 12 weeks
Number of Participants with Adverse Events | up to 12 weeks
  Participants encouraged to contact study staff immediately if they have experienced an adverse event that may or definitely be a result of their involvement in the study. All data collections will include questions on whether the participant believes he/she incurred any possible intervention-related adverse events.

OTHER OUTCOMES:
Improvement in low back pain | up to 12 weeks
  Participants asked to rate how their low back feels compared to when they began treatment on scale 0-6 where 0 is "extremely worsened" and 6 is "extremely improved." Asked at 6 weeks and 12 weeks.
Patient satisfaction | up to 12 weeks
  Satisfaction with treatment of low back pain
Health-related Quality of Life (SF-36) | up to 12 weeks
  The SF-36 is a multi-purpose, generalized health survey that assesses the health benefits produced by a wide range of different treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Saper, MD, MPH, Principal Investigator — Boston Medical Center
Locations (6):
- United States (6):
  - Boston Medical Center, Boston, Massachusetts
  - South Boston Community Health Center, Boston, Massachusetts
  - Dorchester House Multi-service Center, Dorchester, Massachusetts
  - Codman Square Health Center, Dorchester, Massachusetts
  - Upham's Corner Health Center, Dorchester, Massachusetts
  - Roslindale Greater Medical and Dental Center, Roslindale, Massachusetts

REFERENCES:
- [Derived] Cerrada CJ, Weinberg J, Sherman KJ, Saper RB. Inter-method reliability of paper surveys and computer assisted telephone interviews in a randomized controlled trial of yoga for low back pain. BMC Res Notes. 2014 Apr 9;7:227. doi: 10.1186/1756-0500-7-227. PMID 24716775
- [Derived] Saper RB, Boah AR, Keosaian J, Cerrada C, Weinberg J, Sherman KJ. Comparing Once- versus Twice-Weekly Yoga Classes for Chronic Low Back Pain in Predominantly Low Income Minorities: A Randomized Dosing Trial. Evid Based Complement Alternat Med. 2013;2013:658030. doi: 10.1155/2013/658030. Epub 2013 Jun 26. PMID 23878604